CLINICAL TRIAL: NCT04556903
Title: Comparative Effects of Modified Constraint Induced Movement Therapy and Bilateral Arm Training on Upper Extremity in Chronic Stroke Patients
Brief Title: Effects of m CIMT and Bilateral Arm Training on Upper Extremity Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00297 Zobia khan
Record Dates: First submitted 2020-09-16; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Stroke
Keywords: Bilateral Arm Training (BAT); Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Each participant will be requested to draw either number one or number two from a box. Number one will be allocated to Group A and number two will be allocated to group B. The A group will receive mCIMT after applying conservative treatment and Group B will receive BAT for 5 days a week for 8 weeks.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral Arm Training (Experimental): Bilateral Arm Training
  Interventions: Combination Product: Bilateral Arm Training
- modified constrained induce movement therapy (Active Comparator): modified constrained induce movement therapy
  Interventions: Combination Product: modified constrained induce movement therapy

INTERVENTIONS:
Combination Product: Bilateral Arm Training — First component of mCIMT will comprise one hour activity and a rest period of five minute given between each ten minutes of task practice. These activities will base on activities of daily living (ADL'S) and I
  Arms: Bilateral Arm Training
Combination Product: modified constrained induce movement therapy — BAT involves in four sessions, each session involve repetitive practice of bilateral tasks for one hour and a rest period of 5 minutes. The tasks are:
  * Block placement- 10minutes
  * Peg targeting- 10 minutes
  * Peg inversion-10miutes
  * Transferring objects- 10minutes
  Arms: modified constrained induce movement therapy

SUMMARY:
To compare and evaluate the effects of Modified Constraint Induced Movement Therapy (mCIMT) & Bilateral Arm Training on upper extremity in chronic stroke patients this study will be conducted

DETAILED DESCRIPTION:
Stroke is the abrupt loss of neurological function, due to disturbance of the blood flow in the brain. There is variety of crucial sign and symptoms that can occur during stroke include changes in the level of consciousness and impairments of sensation and motor or cognitive function loss. It also includes changes in perceptual and language functions. Worldwide, 55 million people died of stroke in 2002, and approximately 20 percent of these deaths occurred in South Asia. Predicting amounts of deaths from stroke will increase to 63 million in 2015 and 78 million by 2030 with the mass occurring in the poor countries of the world. Rehabilitation plays a major role in minimizing activity limitation and participation restriction or to decrease extent of impairments. Stroke can cause variety of impairments which have greater impact on the patient quality of life. Hemiparesis is the common impairment, in which involvement of upper limb is commonly seen.

mCIMT and BAT techniques both play an important role in the treatment of stroke. In this research, both techniques will be use to evaluate which treatment technique is better for upper extremity chronic stroke patients. Written informed consent will be taken. Each participant will be requested to draw either number one or number two from a box. Number one will be allocated to Group A and number two will be allocated to group B. The A group will receive mCIMT after applying conservative management and Group B will receive BAT for 5 days a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ability to follow instruction & 2 steps command(Mini mental state score > 22)
* At least 6 month after stroke

Exclusion Criteria:

* Spasticity, defined as a score of 3 or more on Modified As worth scale (MAS)
* Uncontrolled hypertension (190/110 mm Hg)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Action Research arm test | 1 hour
  The Action Research Arm Test (ARAT) is a 19 item observational measure used by physical therapists and other health care professionals to assess upper extremity performance (coordination, dexterity and functioning) in stroke recovery,
Fugl-Meyer assessment test (Upper Extremity Section) | 1 hour
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based ... of three evidence based strategies to increase upper extremity function

CONTACTS AND LOCATIONS:
Overall Officials: Zeest Hashmi, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonita R, Beaglehole R. Stroke prevention in poor countries: time for action. Stroke. 2007 Nov;38(11):2871-2. doi: 10.1161/STROKEAHA.107.504589. Epub 2007 Oct 22. No abstract available. PMID 17954904
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] Andrews K, Stewart J. Stroke recovery: he can but does he? Rheumatol Rehabil. 1979 Feb;18(1):43-8. doi: 10.1093/rheumatology/18.1.43. No abstract available. PMID 424667
- [Background] Sterr A, Elbert T, Berthold I, Kolbel S, Rockstroh B, Taub E. Longer versus shorter daily constraint-induced movement therapy of chronic hemiparesis: an exploratory study. Arch Phys Med Rehabil. 2002 Oct;83(10):1374-7. doi: 10.1053/apmr.2002.35108. PMID 12370871
- [Background] Stewart KC, Cauraugh JH, Summers JJ. Bilateral movement training and stroke rehabilitation: a systematic review and meta-analysis. J Neurol Sci. 2006 May 15;244(1-2):89-95. doi: 10.1016/j.jns.2006.01.005. Epub 2006 Feb 14. PMID 16476449
- [Background] Dobkin BH. Clinical practice. Rehabilitation after stroke. N Engl J Med. 2005 Apr 21;352(16):1677-84. doi: 10.1056/NEJMcp043511. PMID 15843670
- [Background] Taub E, Miller NE, Novack TA, Cook EW 3rd, Fleming WC, Nepomuceno CS, Connell JS, Crago JE. Technique to improve chronic motor deficit after stroke. Arch Phys Med Rehabil. 1993 Apr;74(4):347-54. PMID 8466415